CLINICAL TRIAL: NCT00294853
Title: MDCT Calcium Score of Heart Transplanted Patients
Brief Title: Multi Detector-Row Computed Tomography (MDCT) Calcium Score of Heart Transplanted Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-05099
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary calcium score; Coronary artery disease; Cardiac transplantation; Coronary calcium score in heart transplanted patients; Coronary artery disease in heart transplanted patients
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: MDCT calcium score

SUMMARY:
The purpose of the study is to determine if calcium score can be used as a predictor of coronary artery disease in heart transplanted patients, as it is used in non-transplanted persons.

DETAILED DESCRIPTION:
Several studies have shown that a negative calcium score is a strong independent negative predictor of coronary artery disease (CAD). CAD in heart transplants (HTx) differs from CAD lesions in native hearts. The aim of this study is to see if there is a similar relation between coronary artery calcium and CAD in transplanted hearts as in native hearts.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplanted patient
* Aged 18 or above.

Exclusion Criteria:

* Pregnancy
* Atrial fibrillation
* Severe heart failure New York Heart Association (NYHA) class IV
* Severe pulmonary disease making the patient unable to hold his/her breath for more than 10 seconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-12; Study Completion 2007-06

PRIMARY OUTCOMES:
Calcium score | at the date of examination

SECONDARY OUTCOMES:
Coronary stenoses found on coronary angiography | at the date of examination

CONTACTS AND LOCATIONS:
Overall Officials: Anne Günther, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway